CLINICAL TRIAL: NCT02065479
Title: A Pharmacodynamic Study Comparing Prasugrel Versus Ticagrelor in Patients With Coronary Artery Disease Undergoing PCI With CYP2C19 Loss-of-function Genotypes: A Feasibility Study With Point-of-care Pharmacodynamic and Genetic Testing
Brief Title: A Pharmacodynamic Study Comparing Prasugrel Versus Ticagrelor in Patients Undergoing PCI With CYP2C19 Loss-of-function:
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFJ 2014-12; IRB201702750 (Other: UF IRB)
Record Dates: First submitted 2014-02-12; First posted 2014-02-19 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Percutaneous Coronary Intervention; Genetic Polymorphism; Pharmacodynamic
MeSH Terms: conditions — Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Active Comparator): The primary endpoint is the non-inferiority in platelet reactivity of prasugrel versus ticagrelor among CYP2C19 loss of function allele carriers.
  Interventions: Drug: Prasugrel
- Prasugrel (Experimental): The primary endpoint is the non-inferiority in platelet reactivity of prasugrel versus ticagrelor among CYP2C19 loss of function allele carriers.
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Prasugrel — Comparison of platelet reactivity between prasugrel and ticagrelor
  Other Names: Effient
  Arms: Ticagrelor
Drug: Ticagrelor — Comparison of platelet reactivity between prasugrel and ticagrelor
  Other Names: Brilinta
  Arms: Prasugrel

SUMMARY:
Numerous studies have shown that pharmacodynamics (PD) response profiles vary among clopidogrel treated patients and that individuals with reduced response have an increased risk of recurrent ischemic events. There are multiple factors contributing to clopidogrel response variability, including genetic variations of the cytochrome P450 (CYP) 2C19 enzyme. In particular, loss-of-function (LOF) alleles of the CYP2C19 enzyme reduce transformation of clopidogrel pro-drug into its active metabolite. Thus, patients carrying LOF alleles have lower levels of clopidogrel's active metabolite as well as diminished platelet inhibition, which translates into an increased rate of adverse cardiovascular events, particularly in the setting of percutaneous coronary intervention (PCI). Prasugrel and ticagrelor are novel generation P2Y12 receptor inhibitors characterized by greater PD potency and reduced ischemic event rates compared with clopidogrel, and are not affected by CYP2C19 LOF polymorphisms. However, to date there are limited head-to-head PD comparisons between these two new P2Y12 receptors blockers, and there are no studies assessing on how these agents behave among CYP2C19 LOF carriers. The aim of the present study is to compare the PD effects of prasugrel versus ticagrelor in patients undergoing PCI with CYP2C19 LOF alleles using the novel point-of-care genetic testing Spartan RX-CYP2C19 which permits accurate and rapid identification of CYP2C19 genetic status.

DETAILED DESCRIPTION:
Clopidogrel is the most broadly utilized platelet P2Y12 receptor inhibitor. However, numerous studies have shown that pharmacodynamics (PD) response profiles vary among clopidogrel treated patients and that individuals with reduced response have an increased risk of recurrent ischemic events. There are multiple factors contributing to clopidogrel response variability. Among these, genetic variations of the cytochrome P450 (CYP) 2C19 enzyme, a key contributor to clopidogrel metabolism, have been involved. In particular, loss-of-function (LOF) alleles of the CYP2C19 enzyme reduce transformation of clopidogrel pro-drug into its active metabolite. Thus, patients carrying LOF alleles have lower levels of clopidogrel's active metabolite as well as diminished platelet inhibition, which translates into an increased rate of adverse cardiovascular events, particularly in the setting of percutaneous coronary intervention (PCI). Because of these findings, drug regulating authorities have provided a boxed warning on the product label of clopidogrel on the potential for reduced efficacy of clopidogrel among CYP2C19 LOF carriers and suggested considering alternative antiplatelet therapies for these individuals. Prasugrel and ticagrelor are novel generation P2Y12 receptor inhibitors characterized by greater PD potency and reduced ischemic event rates compared with clopidogrel, and are not affected by CYP2C19 LOF polymorphisms. However, to date there are limited head-to-head PD comparisons between these two new P2Y12 receptors blockers, and there are no studies assessing on how these agents behave among CYP2C19 LOF carriers. Tailoring antiplatelet therapy according to results of genetic testing has been limited in real world clinical practice because of not having readily accessible results of individual's genetic makeup. The aim of the present study is to compare the PD effects of prasugrel versus ticagrelor in patients undergoing PCI with CYP2C19 LOF alleles using the novel point-of-care genetic testing Spartan RX-CYP2C19 which permits accurate and rapid identification of CYP2C19 genetic status.

ELIGIBILITY:
* Inclusion criteria:

  1. Patients scheduled for left heart catheterization and undergoing PCI
  2. Age 18-75 years
  3. On aspirin (81mg) or aspirin (81mg) and clopidogrel (75mg/day)
  4. Presence of at least one 2C19 LOF allele
* Exclusion criteria:

  1. Known allergies to aspirin, prasugrel, ticagrelor, or clopidogrel
  2. Age >75 years
  3. Weight <60kg
  4. Considered at high risk for bleeding
  5. History of ischemic or hemorrhagic stroke or transient ischemic attack
  6. Known severe hepatic dysfunction
  7. On treatment with oral anticoagulant therapy (Vitamin K antagonists, dabigatran, apixaban, rivaroxaban)
  8. Use of glycoprotein IIb/IIIa inhibitors (abciximab, eptifibatide, tirofiban)
  9. Blood dyscrasia or bleeding diathesis
  10. Platelet count <80x106/mL
  11. Hemoglobin <10 g/dL.
  12. Active bleeding or hemodynamic instability
  13. Creatinine Clearance <30 mL/minute
  14. Patients with sick sinus syndrome (SSS) or high degree AV block without pacemaker protection.
  15. Current treatment with drugs interfering with CYP3A4 metabolism (to avoid interaction with Ticagrelor): Ketoconazole, itraconazole, voriconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, and telithromizycin.
  16. Pregnant females* *Women of childbearing age must use reliable birth control (i.e. oral contraceptives) while participating in the study.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-03; Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franchi F, Rollini F, Rivas J, Rivas A, Agarwal M, Briceno M, Wali M, Nawaz A, Silva G, Shaikh Z, Maailiki N, Been L, Pineda AM, Suryadevara S, Soffer D, Zenni MM, Bass TA, Angiolillo DJ. Prasugrel Versus Ticagrelor in Patients With CYP2C19 Loss-of-Function Genotypes: Results of a Randomized Pharmacodynamic Study in a Feasibility Investigation of Rapid Genetic Testing. JACC Basic Transl Sci. 2020 Mar 25;5(5):419-428. doi: 10.1016/j.jacbts.2020.02.009. eCollection 2020 May. PMID 32478205

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ticagrelor | Prasugrel
Started | 33 | 32
Completed | 33 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor | Prasugrel | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (8) | 60 (9) | 59 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 26 | 25 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 23 | 21 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 32 | 65
Diabetes Mellitus [Count of Participants; unit: Participants] | 10 | 14 | 24

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity
Description: The primary endpoint is P2Y12 reaction unit (PRU) measured by the Verify Now P2Y12 assay 24hours/hospital discharge post randomization to prasugrel vs ticagrelor. PRU is is an arbitrary unit of measure to assess ADP-induced platelet aggregation.
Time Frame: 24 hours post loading dose
Measure: Mean (Standard Deviation); unit: PRU
Arm/Group | Ticagrelor | Prasugrel
Number analyzed (Participants) | 33 | 32
PRU | 36 (41) | 33 (56)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Ticagrelor | Prasugrel
All-Cause Mortality (participants affected / at risk) | 33/33 | 32/32
Serious Adverse Events (participants affected / at risk) | 0/33 | 1/32
Other Adverse Events (participants affected / at risk) | 3/33 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor (N=33) | Prasugrel (N=32)
Stroke (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor (N=33) | Prasugrel (N=32)
Dypnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT02065479/Prot_SAP_000.pdf